CLINICAL TRIAL: NCT03273517
Title: Caregivers and Resident Doctors' Perceptions of Preoperative Fasting in Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Faculdade de Ciências Médicas da Santa Casa de São Paulo (Other)
Responsible Party: Principal Investigator, Lígia Andrade da Silva Telles mathias, Doctor, Faculdade de Ciências Médicas da Santa Casa de São Paulo
Other Study IDs: 58080016.8.0000.5472
Record Dates: First submitted 2017-06-29; First posted 2017-09-06 (Actual); Last update posted 2017-09-06 (Actual); Status verified 2017-06

CONDITIONS: Fasting
Keywords: Glycemia; Preoperative fasting; Pediatric patients; Anesthesia; Knowledge of the resident
MeSH Terms: conditions — Fasting | interventions — Elective Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Elective surgery — Elective surgery in children aged 0-15 years ASA I and II

SUMMARY:
Historically, adults and children who undergo elective surgery remain fasting in the preoperative period, for the purposes of avoiding bronchial aspiration of the gastric contents during general anesthesia. The determination of preoperative fasting has taken on importance only in 1946, when Mendelson established a relationship between pulmonary aspiration during labor and general anesthesia. Stemming from other studies, such concept has been expanded to elective surgery and 25 ml were set as the maximum threshold of the gastric content to thus reduce the hazards of aspiration pneumonia.

The fasting time prescribed is still the subject of several investigations. For decades it has been established that patients should not feed on solids or ingest liquids over a period of 8 to 12 hours prior to surgery.

The guidelines are well set in connection with the rules of fasting, with aims at making the instructions constant throughout different services worldwide. In 2011, the American and the European guidelines became more permissive and determined as safe the 2 hours for liquids devoid of residue, 4 hours for breast milk, 6 hours for infant formula and non-human milk, 6 hours for light meals, and 8 hours for full meals. In accordance with the American guideline, liquids devoid of residue are: water, fruit juice with no pulp, carbohydrate-based beverages, tea with no residue, and black coffee, but those examples are not extensive. Gelatin is solid prior to intake, but it is found in a liquid state inside the stomach and, therefore, it is regarded as a liquid devoid of residue. Yet, in spite of the non-human milk's being a liquid material, it features a gastric emptying time which is similar to that of the non-fat solids. A light meal is characterized by toast and liquids devoid of residue, whilst a full meal includes food that is fried or which contains a high level of fat.

Currently, many directives (American Society of Anaesthesiologists - ASA; Norwegian National Consensus Guideline - NNCG; Association of Anaesthetists of Great Britain and Ireland - AAGBI) recommend liquids devoid of residue until two hours prior to the anesthetic induction for elective surgery in healthy children. The particular benefit of the oral intake of fluids includes a lower incidence of deleterious effects, such as thirst, irritation, crying, hypoglycemia, and dehydration. The preservation of the intravascular volume improves the hemodynamic conditions during the induction of inhalation anesthesia and facilitates the vascular access.

Even though the old instruction of "nothing by mouth after midnight" is in a process of being replaced by shorter periods of fasting, both surgeons and anesthesiologists still deem the traditional fast indispensable and have trouble with implementing the new norms, either by uncertainty before the possibility of the catastrophic consequences of pulmonary aspiration, or by lack of update on the subject. That matter generates mistakes in the rendering of information by the health professionals. Combined with the unawareness of the guardians in respect of the risk of bronchial aspiration and the anxiety in relation to the fasting, there is a result of difficulty in abidance by the proper preoperative fasting.

The minority of the guardians understands the real importance of the preoperative fasting and, many times, food regarded as "harmless" is offered during the period of fasting. Likewise, the guardians provide improper information in order to maintain the surgical procedure, with no regard for the correct observance of the fasting. That way, countless pediatric elective surgeries are canceled, deriving in psychological, social, and economic implications. The correction of these flaws will allow for the anesthetic procedure to take place in a more secure manner, with the proper observance of the fasting period and with the least possible trauma to the child.

DETAILED DESCRIPTION:
Cross-sectional, observational study in which questionnaires will be applied to the guardians during the immediate post-surgical period in the anesthetic recovery room by residents of the third year of anesthesiology.

Moreover, the knowledge of the physicians of the surgical specialties of the aforementioned institution pursuant to preoperative fasting is to be assessed, whilst a questionnaire will be applied after the meetings of the respective departments.

After explication of the study, the Informed Consent Form will be handed in the pre-anesthetic consultation, and the questionnaires will be applied in the post-anesthetic recovery room to the guardians of the children who have undergone imaging examination and elective surgery. After the anesthetic induction, the patients will be subject to the measurement of blood glucose by Dextro. The resident doctors will be evaluated by means of another questionnaire, which is to be applied after the weekly clinical meeting of each specialty.

ELIGIBILITY:
Inclusion Criteria:

* Literate parents or guardians;
* Children with indication for general anesthesia;
* Children between 0 and 15 years of age;
* Children with ASA I and II physical condition.
* Resident doctors of the specialties of general and pediatric surgery, ophthalmology, otorhinolaryngology, anesthesia, general orthopedics, a pediatric orthopedics.

Exclusion Criteria:

* Children subject to anesthetic induction by means of the rapid sequence technique.
* Children with alterations in the gastric emptying (diabetes, obesity, neonatal hypoxic encephalopathy, usage of gastrostomy and of nasogastric and nasoenteric probes).

Max Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: * Children below 15 years of age, subject to ophthalmological, otorhinolaryngological, orthopedic, and pediatric elective surgery and imaging examinations, with ASA I and II physical condition, and their guardians, over a period of three months.
  * Resident doctors of the specialties of general and pediatric surgery, ophthalmology, otorhinolaryngology, anesthesia, general orthopedics, a pediatric orthopedics.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-11-01 (Estimated)

PRIMARY OUTCOMES:
Glycemia | An average of 1 hour after induction of general anesthesia
  After the anesthetic induction, the patients will be subject to the measurement of blood glucose by Dextro.
The understanding and the perception of the guardians in relation to the importance of fasting in pediatric patients | 1 hour after post-anesthetic
  The questionnaires will be applied to the guardians of the children who have undergone imaging examination and elective surgery

SECONDARY OUTCOMES:
Knowledge of the resident doctors | Through study completion, an average of 1 year
  The knowledge of the physicians of the surgical specialties of the aforementioned institution pursuant to preoperative fasting is to be assessed, whilst a questionnaire will be applied

CONTACTS AND LOCATIONS:
Locations (1):
- Santa Casa of São Paulo Medical School, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Buller Y, Sims C. Prolonged fasting of children before anaesthesia is common in private practice. Anaesth Intensive Care. 2016 Jan;44(1):107-10. doi: 10.1177/0310057X1604400116. PMID 26673596
- [Result] Cantellow S, Lightfoot J, Bould H, Beringer R. Parents' understanding of and compliance with fasting instruction for pediatric day case surgery. Paediatr Anaesth. 2012 Sep;22(9):897-900. doi: 10.1111/j.1460-9592.2012.03903.x. Epub 2012 Jun 25. PMID 22731386
- [Result] Cook-Sather SD, Litman RS. Modern fasting guidelines in children. Best Pract Res Clin Anaesthesiol. 2006 Sep;20(3):471-81. doi: 10.1016/j.bpa.2006.02.003. PMID 17080697
- [Result] Flick RP, Schears GJ, Warner MA. Aspiration in pediatric anesthesia: is there a higher incidence compared with adults? Curr Opin Anaesthesiol. 2002 Jun;15(3):323-7. doi: 10.1097/00001503-200206000-00008. PMID 17019220
- [Result] Green CR, Pandit SK, Schork MA. Preoperative fasting time: is the traditional policy changing? Results of a national survey. Anesth Analg. 1996 Jul;83(1):123-8. doi: 10.1097/00000539-199607000-00022. PMID 8659722
- [Result] Kushnir J, Djerassi R, Sofer T, Kushnir T. Threat perception, anxiety and noncompliance with preoperative fasting instructions among mothers of children attending elective same day surgery. J Pediatr Surg. 2015 May;50(5):869-74. doi: 10.1016/j.jpedsurg.2014.08.018. Epub 2014 Oct 1. PMID 25783336
- [Result] MENDELSON CL. The aspiration of stomach contents into the lungs during obstetric anesthesia. Am J Obstet Gynecol. 1946 Aug;52:191-205. doi: 10.1016/s0002-9378(16)39829-5. No abstract available. PMID 20993766
- [Result] Moro ET. [Prevention of pulmonary gastric contents aspiration.]. Rev Bras Anestesiol. 2004 Apr;54(2):261-75. doi: 10.1590/s0034-70942004000200014. Portuguese. PMID 19471734
- [Result] Ramirez-Mora J, Moyao-Garcia D, Nava-Ocampo AA. Attitudes of Mexican anesthesiologists to indicate preoperative fasting periods: A cross-sectional survey. BMC Anesthesiol. 2002 May 17;2(1):3. doi: 10.1186/1471-2253-2-3. PMID 12019024
- [Result] Schreiner MS, Triebwasser A, Keon TP. Ingestion of liquids compared with preoperative fasting in pediatric outpatients. Anesthesiology. 1990 Apr;72(4):593-7. doi: 10.1097/00000542-199004000-00002. PMID 2321772
- [Result] Smith I, Kranke P, Murat I, Smith A, O'Sullivan G, Soreide E, Spies C, in't Veld B; European Society of Anaesthesiology. Perioperative fasting in adults and children: guidelines from the European Society of Anaesthesiology. Eur J Anaesthesiol. 2011 Aug;28(8):556-69. doi: 10.1097/EJA.0b013e3283495ba1. PMID 21712716
- [Result] Warner MA. Is pulmonary aspiration still an important problem in anesthesia? Curr Opin Anaesthesiol. 2000 Apr;13(2):215-8. doi: 10.1097/00001503-200004000-00023. PMID 17016306
- [Result] American Society of Anesthesiologists Committee. Practice guidelines for preoperative fasting and the use of pharmacologic agents to reduce the risk of pulmonary aspiration: application to healthy patients undergoing elective procedures: an updated report by the American Society of Anesthesiologists Committee on Standards and Practice Parameters. Anesthesiology. 2011 Mar;114(3):495-511. doi: 10.1097/ALN.0b013e3181fcbfd9. No abstract available. PMID 21307770